CLINICAL TRIAL: NCT04616027
Title: A PHASE 1, OPEN-LABEL, SINGLE-DOSE, PARALLEL GROUP STUDY TO EVALUATE THE PHARMACOKINETICS OF PF-06882961 IN PARTICIPANTS WITH TYPE 2 DIABETES MELLITUS WITH VARYING DEGREES OF RENAL IMPAIRMENT RELATIVE TO PARTICIPANTS WITHOUT RENAL IMPAIRMENT
Brief Title: STUDY OF PF-06882961 IN PARTICIPANTS WITH TYPE 2 DIABETES MELLITUS WITH VARYING DEGREES OF RENAL IMPAIRMENT AND PARTICIPANTS WITHOUT RENAL IMPAIRMENT
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: C3421012
Record Dates: First submitted 2020-10-29; First posted 2020-11-04 (Actual); Results first posted 2024-05-10 (Actual); Last update posted 2024-05-10 (Actual); Status verified 2023-12

CONDITIONS: Diabetes Mellitus, Type 2; Renal Impairment; Healthy
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Renal Insufficiency | interventions — danuglipron

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Healthy participants with normal renal function (Experimental): This arm includes participants with normal renal function who will receive an oral dose of PF-06882961 20 milligrams (mg) on Day 1
  Interventions: Drug: PF-06882961 20 mg
- Participants with T2DM with normal renal function (Experimental): This arm includes participants with Type 2 Diabetes Mellitus (T2DM) with normal renal function who will receive an oral dose of PF-06882961 20 mg on Day 1
  Interventions: Drug: PF-06882961 20 mg
- Participants with T2DM with mild renal impairment (Experimental): This arm includes participants with Type 2 Diabetes Mellitus (T2DM) with mild renal impairment who will receive an oral dose of PF-06882961 20 mg on Day 1
  Interventions: Drug: PF-06882961 20 mg
- Participants with T2DM with moderate renal impairment (Experimental): This arm includes participants with Type 2 Diabetes Mellitus (T2DM) with moderate renal impairment who will receive an oral dose of PF-06882961 20 mg on Day 1
  Interventions: Drug: PF-06882961 20 mg
- Participants with T2DM with severe renal impairment (Experimental): This arm includes participants with Type 2 Diabetes Mellitus (T2DM) with severe renal impairment who will receive an oral dose of PF-06882961 20 mg on Day 1
  Interventions: Drug: PF-06882961 20 mg

INTERVENTIONS:
Drug: PF-06882961 20 mg — PF-06882961 20 mg single oral dose provided in tablet form administered in a fed state on Day 1

SUMMARY:
This study will characterize the effect of varying degrees of renal impairment on the pharmacokinetics (PK), safety and tolerability of a single oral dose of PF- 06882961 compared with participants with normal renal function.

ELIGIBILITY:
Inclusion Criteria:

* Stable renal function (for participants not on dialysis) defined as ≤25% difference between 2 measurements of eGFR (as calculated by the sponsor-identified central laboratory using the CKD-EPI equation)1 obtained at Screening visits S1 and S2. The average of the 2 eGFR values obtained from S1 and S2 will be used for study enrollment and assignment to appropriate renal function group. Note: participants on dialysis will be placed in Group 5 regardless of eGFR from S1 and S2 (S2 is optional for dialysis participants only).
* Male and female participants must be ≥18 years of age, inclusive, at the time of signing the informed consent document (ICD).
* Participants who are willing and able to comply with all scheduled visits, treatment plan, laboratory tests, lifestyle considerations, and other study procedures, including the ability to perform self-monitoring blood glucose at a frequency deemed appropriate by the investigator.
* Body mass index (BMI) of ≥18.0 kg/m2 and <45.4 kg/m2; and a total body weight >50 kg (110 lb).
* Capable of giving signed informed consent, which includes compliance with the requirements and restrictions listed in the ICD and in this protocol.

Additional Inclusion Criteria for Healthy Participants with Normal Renal

Function (Group 1):

* No clinically relevant abnormalities identified by a detailed medical history, full physical examination, including blood pressure (BP) and pulse rate measurement, standard 12-lead ECG and clinical laboratory tests.
* Normal renal function (mean eGFR ≥90 mL/min) based on an average of measures from Screening visits S1 and S2.
* Demographically comparable to participants with impaired renal function:

  1. A body weight within ±15 kg of the mean body weight of the pooled renal impairment groups (Groups 3, 4, and 5), as provided by sponsor;
  2. An age within ±10 years of the mean age of the pooled renal impairment groups (Groups 3, 4 and 5), as provided by sponsor;
  3. Attempts will be made to ensure that the male to female distribution in Group 1 is comparable to that in the pooled renal impairment groups (Cohorts 3, 4, and 5).

     Additional Inclusion Criteria for T2DM Participants with Normal Renal

     Function (Group 2):
* A prior diagnosis of T2DM with an HbA1c ≥6% and ≤10.5%, at Screening visit S1, confirmed by a single repeat, if deemed necessary.
* Normal renal function (mean eGFR ≥90 mL/min) based on an average of measures from Screening visits S1 and S2.
* Prohibited prior/concomitant medications.
* Demographically comparable to participants with impaired renal function:

  1. A body weight within ±15 kg of the mean body weight of the pooled renal impairment groups (Groups 3, 4, and 5), as provided by sponsor;
  2. An age within ±10 years of the mean age of the pooled renal impairment groups (Groups 3, 4, and 5), as provided by sponsor;
  3. Attempts will be made to ensure that the male to female distribution in Group 2 is comparable to that in the pooled renal impairment groups (Cohorts 3, 4, and 5).

Additional Inclusion Criteria for T2DM Participants with Impaired Renal Function (Groups 3-5):

* A prior diagnosis of T2DM with an HbA1c ≥6% and ≤10.5%, at Screening visit S1, confirmed by a single repeat, if deemed necessary.
* Meet the eGFR criteria listed for Groups 3, 4, or 5 (for participants not on dialysis) in Table 1 based on an average of measures from Screening visits S1 and S2.
* Stable concomitant medications, as defined in Section 6.5, for the management of medical conditions relevant to an individual participant's medical history. Participants receiving fluctuating concomitant medications/treatments may be considered, on a case-by-case basis with input from sponsor, if the underlying disease is stable.
* For Group 5 participants on dialysis only, participants must have required hemodialysis for at least 6 weeks and need dialysis sessions 3 times per week

Exclusion Criteria:

* Other acute or chronic medical or psychiatric condition including recent (within the past year) or active suicidal ideation or behavior or laboratory abnormality that may increase the risk associated with study participation or IP administration or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the participant inappropriate for entry into this study.
* Any condition possibly affecting drug absorption (eg, prior bariatric surgery, gastrectomy, or any area of intestinal resection, active inflammatory bowel disease or pancreatic insufficiency). NOTE: subjects who have undergone cholecystectomy and/or appendectomy are eligible for this study so long as the surgery occurred more than 6 months prior to Screening;
* Any malignancy not considered cured (except basal cell carcinoma and squamous cell carcinoma of the skin); a participant is considered cured if there has been no evidence of cancer recurrence in the previous 5 years.
* Personal or family history of medullary thyroid carcinoma (MTC) or multiple endocrine neoplasia syndrome type 2 (MEN2), or participants with suspected MTC per the investigator's judgement.
* History of chronic or acute pancreatitis within 5 years.
* Diagnosis of type 1 diabetes mellitus or secondary forms of diabetes.
* History of diabetic ketoacidosis.
* History of myocardial infarction, unstable angina, arterial revascularization, stroke, New York Heart Association Functional Class II-IV heart failure, or transient ischemic attack within 3 months of Screening visit S1.
* Urinary incontinence.
* Participants with acute renal disease.
* Renal allograft recipients.
* Participants with other clinically significant disease, in the judgment of the investigator that may affect the safety of the participant or that may affect the PK of PF 06882961.
* Prohibited prior/concomitant medications.
* Compliance with details regarding prohibited prior/concomitant medications.
* Previous administration with an investigational drug within 30 days (or as determined by the local requirement) or 5 half-lives preceding the first dose of IP used in this study (whichever is longer).
* Known prior participation in a trial involving PF 06882961 or known hypersensitivity or intolerance to a GLP-1R agonist.
* Screening standard 12-lead ECG that demonstrates a clinically relevant abnormality that requires further diagnostic evaluation or intervention (eg, new, clinically relevant arrhythmia, conduction disturbance, findings suggestive of ischemia). A potential participant whose pre-dose ECG (on Day 1, 0 hour) demonstrates a clinically relevant abnormality that requires further diagnostic evaluation or intervention will be considered a screen failure.
* A positive COVID-19 test in the screening period.
* A positive urine drug test (or other type of drug test in anuric participants on dialysis only).
* Participants with ANY of the following abnormalities in clinical laboratory tests at Screening, as assessed by the study specific central laboratory and confirmed by a single repeat test, if deemed necessary:

  • Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) level ≥2 × upper limit of normal (ULN);
  * Total bilirubin level ≥1.5 × ULN; participants with a history of Gilbert's syndrome may have direct bilirubin measured and would be eligible for this study provided the direct bilirubin level is ≤ ULN.
  * Fasting C-peptide <0.8 ng/mL.
  * Fasting plasma glucose (FPG) >270 mg/dL (15 mmol/L) at screening (S1).
* History of regular alcohol consumption exceeding 7 drinks/week for female participants or 14 drinks/week for male participants (1 drink = 5 ounces [150 mL] of wine or 12 ounces [360 mL] of beer or 1.5 ounces [45 mL] of hard liquor) within 6 months before screening.
* Blood donation (excluding plasma donations) of approximately 1 pint (500 mL) or more within 60 days prior to dosing.
* History of sensitivity to heparin or heparin-induced thrombocytopenia only if heparin is planned to flush intravenous catheters.

Additional Exclusion Criteria for Healthy Participants with Normal Renal

Function (Group 1):

- Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic, or allergic disease (including clinically relevant and significant drug allergies, but excluding untreated, asymptomatic, seasonal allergies at time of dosing).

* Use of prescription or non-prescription drugs and dietary and herbal supplements within 14 days or 5 half-lives (whichever is longer) prior to the first dose of IP). As an exception, ibuprofen or acetaminophen may be used at doses of ≤1 g/day. Limited use of non-prescription medications that are not believed to affect participant safety or the overall results of the study may be permitted on a case-by-case basis following approval by the sponsor.
* Screening seated systolic blood pressure (SBP) >140 mmHg or diastolic blood pressure (DBP) >90 mmHg, following at least 5 minutes of supine rest. If SBP is >140 mmHg or DBP >90 mmHg, the BP should be repeated 2 more times and the average of the 3 BP values should be used to determine the participant's eligibility.
* Participants with ANY of the following abnormalities in clinical laboratory tests at Screening, as assessed by the study specific central laboratory and confirmed by a single repeat test, if deemed necessary:

HbA1c ≥6.0% at Screening visit S1; FPG ≥126 mg/dL at screening (S1); Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) level ≥1.5 × upper limit of normal (ULN). Additional Exclusion Criteria for T2DM Participants with Normal Renal

Function (Group 2):

- At Screening, seated systolic blood pressure (SBP) ≥160 mm Hg and/or diastolic blood pressure (DBP) ≥105 mm Hg after ≥5minute of seated rest, with a single repeat permitted to assess eligibility, if needed, at each of these 2 visits.

Additional Exclusion Criteria for T2DM Participants with Impaired Renal

Function (Groups 3-5) only:

- At Screening, persistent severe, uncontrolled hypertension; for example: seated systolic blood pressure (SBP) ≥180 mm Hg and/or diastolic blood pressure (DBP) ≥105 mm Hg after ≥5minute of seated rest, with a single repeat permitted to assess eligibility, if needed, at each of these 2 visits: For subjects with SBP ≥160 mm Hg or DBP ≥100 mm Hg, the period between Screening and Day 1 must be used to refine the doses of the agents used for management of blood pressure with the aim to have stable BP on Day 1;.

- For participants in Group 5 on Dialysis only: Hemodynamic instability during or at the conclusion of dialysis during the 2 weeks prior to dosing, as marked by symptomatic hypotension.

Criteria for Dosing on Day 1

Participants will progress to dosing on Day 1 provided they have satisfied all the following criteria:

* In women of childbearing potential, urine pregnancy test on Day -1 is negative;
* Cohort 1 and Cohort 2 only: Approval from the sponsor must be obtained before proceeding with dosing participants in either Cohort 1 or Cohort 2;
* Cohorts 2-5 only: Participants must have measurement on Day 1 of SBP <160 mm Hg and DBP <100 mm Hg; A single repeat assessment is permitted, to confirm that the above criterion is met [and in such cases, the repeat assessment overrides initial results].

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2021-01-13 (Actual); Primary Completion 2022-02-18 (Actual); Study Completion 2022-02-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (3):
- United States (3):
  - University of Miami Hospital, Miami, Florida
  - Orlando Clinical Research Center, Orlando, Florida
  - Prism Research LLC dba Nucleus Network, Saint Paul, Minnesota

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- [Derived] Fediuk DJ, Gorman DN, Stoddard SA, Zhang Y, Ogden AG, Winton JA, Saxena AR. Effect of Renal Impairment on the Pharmacokinetics of a Single Oral Dose of Danuglipron in Participants With Type 2 Diabetes. J Clin Pharmacol. 2024 Apr;64(4):449-460. doi: 10.1002/jcph.2371. Epub 2023 Nov 2. PMID 37840155
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C3421012

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants were allocated to treatment at 3 sites in 1 country. 42 participants were allocated to treatment, 3 did not receive treatment. A total of 39 participants were treated and completed the study.
Groups:
- Healthy and Normal Renal Function: Healthy participants whose estimated glomerular filtration rate (eGFR) ≥90mL/min were included in this group. PF-06882961 was administered at a dose of 20 mg on Day 1.
- T2DM Normal Renal Function: Participants with type 2 diabetes mellitus (T2DM) whose estimated glomerular filtration rate (eGFR) ≥90mL/min were included in this group. PF-06882961 was administered at a dose of 20 mg on Day 1.
- T2DM Mild Renal Impairment: Participants with T2DM whose estimated glomerular filtration rate (eGFR) 60-89mL/min were included in this group. PF-06882961 was administered at a dose of 20 mg on Day 1.
- T2DM Moderate Renal Impairment: Participants with T2DM whose estimated glomerular filtration rate (eGFR) 30-59mL/min were included in this group. PF-06882961 was administered at a dose of 20 mg on Day 1.
- T2DM Severe Renal Impairment: Participants with T2DM whose estimated glomerular filtration rate (eGFR) <30mL/min were included in this group. PF-06882961 was administered at a dose of 20 mg on Day 1.
Period: Overall Study
Arm/Group | Healthy and Normal Renal Function | T2DM Normal Renal Function | T2DM Mild Renal Impairment | T2DM Moderate Renal Impairment | T2DM Severe Renal Impairment
Started | 8 | 7 | 8 | 8 | 8
Completed | 8 | 7 | 8 | 8 | 8
Not Completed | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All enrolled participants who received at least one dose of study intervention.
Groups:
- Total: Total of all reporting groups
Arm/Group | Healthy and Normal Renal Function | T2DM Normal Renal Function | T2DM Mild Renal Impairment | T2DM Moderate Renal Impairment | T2DM Severe Renal Impairment | Total
Number analyzed (Participants) | 8 | 7 | 8 | 8 | 8 | 39
Age, Continuous [Mean (Standard Deviation); unit: Years] | 57.1 (2.30) | 64.1 (7.17) | 68.0 (10.90) | 67.0 (9.09) | 59.8 (4.98) | 63.2 (8.31)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 4 | 5 | 4 | 2 | 18
  Male | 5 | 3 | 3 | 4 | 6 | 21
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 0 | 2 | 3 | 4 | 14
  Not Hispanic or Latino | 3 | 7 | 6 | 5 | 4 | 25
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 6 | 4 | 7 | 7 | 4 | 28
  Black or African American | 1 | 3 | 1 | 1 | 4 | 10
  American Indian or Alaska Native | 1 | 0 | 0 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Maximum Observed Plasma Concentration (Cmax) of Plasma PF-06882961
Description: Cmax was the maximum observed plasma concentration and was directly observed from data.
Time Frame: 0 (pre dose), 1, 2, 3, 4, 5, 6, 8, 10, 12, 16 hours (post dose) on Day 1, 24 and 36 hours (post dose) on Day 2, 48 hours (post dose) on Day 3
Population: All participants who received at least 1 dose of PF-06882961 and had at least 1 of the plasma PK parameters of interest calculated. Here, overall number of participants analyzed signifies number of participants evaluable for this outcome measure.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms/milliliter (ng/mL)
Arm/Group | Healthy and Normal Renal Function | T2DM Normal Renal Function | T2DM Mild Renal Impairment | T2DM Moderate Renal Impairment | T2DM Severe Renal Impairment
Number analyzed (Participants) | 8 | 7 | 7 | 8 | 8
nanograms/milliliter (ng/mL) | 38.80 (28) | 38.67 (58) | 39.19 (42) | 56.68 (28) | 39.18 (50)
Statistical Analysis 1: Comparison: Healthy and Normal Renal Function vs T2DM Normal Renal Function; "T2DM Normal Renal Function" was test, "Healthy and Normal Renal Function" was reference; Test type: Other — ANOVA; Ratio (Test/Reference) of Adjusted Means = 99.67, 90% CI 2-sided [70.15 to 141.60]
Statistical Analysis 2: Comparison: T2DM Normal Renal Function vs T2DM Mild Renal Impairment; "T2DM Mild Renal Impairment" was test, "T2DM Normal Renal Function" was reference; Test type: Other — ANOVA; Ratio (Test/Reference) of Adjusted Means = 101.34, 90% CI 2-sided [70.51 to 145.63]
Statistical Analysis 3: Comparison: T2DM Normal Renal Function vs T2DM Moderate Renal Impairment; "T2DM Moderate Renal Impairment" was test, "T2DM Normal Renal Function" was reference; Test type: Other — ANOVA; Ratio (Test/Reference) of Adjusted Means = 146.56, 90% CI 2-sided [103.16 to 208.22]
Statistical Analysis 4: Comparison: T2DM Normal Renal Function vs T2DM Severe Renal Impairment; "T2DM Severe Renal Impairment" was test, "T2DM Normal Renal Function" was reference; Test type: Other — ANOVA; Ratio (Test/Reference) of Adjusted Means = 101.31, 90% CI 2-sided [71.31 to 143.92]

2. Primary Outcome: Area Under the Plasma Concentration-Time Profile From Time Zero Extrapolated to Infinite Time (AUCinf) of Plasma PF-06882961
Description: AUCinf was defined as area under the plasma concentration-time curve from time zero to infinity.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms*hour/milliliter (ng*hr/mL)
Arm/Group | Healthy and Normal Renal Function | T2DM Normal Renal Function | T2DM Mild Renal Impairment | T2DM Moderate Renal Impairment | T2DM Severe Renal Impairment
Number analyzed (Participants) | 8 | 7 | 6 | 7 | 8
nanograms*hour/milliliter (ng*hr/mL) | 362.4 (30) | 404.8 (49) | 487.0 (19) | 543.2 (48) | 408.8 (46)
Statistical Analysis 1: Comparison: Healthy and Normal Renal Function vs T2DM Normal Renal Function; "T2DM Normal Renal Function" was test, "Healthy and Normal Renal Function" was reference; Test type: Other — ANOVA; Ratio (Test/Reference) of Adjusted Means = 111.71, 90% CI 2-sided [79.52 to 156.93]
Statistical Analysis 2: Comparison: T2DM Normal Renal Function vs T2DM Mild Renal Impairment; "T2DM Mild Renal Impairment" was test, "T2DM Normal Renal Function" was reference; Test type: Other — ANOVA; Ratio (Test/Reference) of Adjusted Means = 120.31, 90% CI 2-sided [83.49 to 173.38]
Statistical Analysis 3: Comparison: T2DM Normal Renal Function vs T2DM Moderate Renal Impairment; "T2DM Moderate Renal Impairment" was test, "T2DM Normal Renal Function" was reference; Test type: Other — ANOVA; Ratio (Test/Reference) of Adjusted Means = 134.18, 90% CI 2-sided [94.46 to 190.62]
Statistical Analysis 4: Comparison: T2DM Normal Renal Function vs T2DM Severe Renal Impairment; "T2DM Severe Renal Impairment" was test, "T2DM Normal Renal Function" was reference; Test type: Other — ANOVA; Ratio (Test/Reference) of Adjusted Means = 100.99, 90% CI 2-sided [71.89 to 141.87]

3. Primary Outcome: Area Under the Plasma Concentration-Time Profile From Time Zero to Time of the Last Quantifiable Concentration (AUClast) of Plasma PF-06882961
Description: AUClast was area under the plasma concentration time-curve from zero (pre-dose) to the last measured concentration.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | Healthy and Normal Renal Function | T2DM Normal Renal Function | T2DM Mild Renal Impairment | T2DM Moderate Renal Impairment | T2DM Severe Renal Impairment
Number analyzed (Participants) | 8 | 7 | 7 | 8 | 8
ng*hr/mL | 359.9 (30) | 399.6 (50) | 466.3 (19) | 538.2 (44) | 404.8 (46)
Statistical Analysis 1: Comparison: Healthy and Normal Renal Function vs T2DM Normal Renal Function; "T2DM Normal Renal Function" was test, "Healthy and Normal Renal Function" was reference; Test type: Other — ANOVA; Ratio (Test/Reference) of Adjusted Means = 111.02, 90% CI 2-sided [79.60 to 154.86]
Statistical Analysis 2: Comparison: T2DM Normal Renal Function vs T2DM Mild Renal Impairment; "T2DM Mild Renal Impairment" was test, "T2DM Normal Renal Function" was reference; Test type: Other — ANOVA; Ratio (Test/Reference) of Adjusted Means = 116.70, 90% CI 2-sided [82.76 to 164.56]
Statistical Analysis 3: Comparison: T2DM Normal Renal Function vs T2DM Moderate Renal Impairment; "T2DM Moderate Renal Impairment" was test, "T2DM Normal Renal Function" was reference; Test type: Other — ANOVA; Ratio (Test/Reference) of Adjusted Means = 134.68, 90% CI 2-sided [96.56 to 187.85]
Statistical Analysis 4: Comparison: T2DM Normal Renal Function vs T2DM Severe Renal Impairment; "T2DM Severe Renal Impairment" was test, "T2DM Normal Renal Function" was reference; Test type: Other — ANOVA; Ratio (Test/Reference) of Adjusted Means = 101.31, 90% CI 2-sided [72.63 to 141.30]

4. Primary Outcome: Fraction Unbound (fu) of Plasma PF-06882961
Description: Fu was defined as fraction of unbound drug in plasma.
Time Frame: 0 (pre dose), 4 hours (post dose) on Day 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio
Arm/Group | Healthy and Normal Renal Function | T2DM Normal Renal Function | T2DM Mild Renal Impairment | T2DM Moderate Renal Impairment | T2DM Severe Renal Impairment
Number analyzed (Participants) | 8 | 7 | 7 | 8 | 8
Ratio | 0.01519 (9) | 0.01542 (15) | 0.01699 (14) | 0.01861 (18) | 0.01960 (18)
Statistical Analysis 1: Comparison: Healthy and Normal Renal Function vs T2DM Normal Renal Function; "T2DM Normal Renal Function" was test, "Healthy and Normal Renal Function" was reference; Test type: Other — ANOVA; Ratio (Test/Reference) of Adjusted Means = 101.52, 90% CI 2-sided [88.89 to 115.94]
Statistical Analysis 2: Comparison: T2DM Normal Renal Function vs T2DM Mild Renal Impairment; "T2DM Mild Renal Impairment" was test, "T2DM Normal Renal Function" was reference; Test type: Other — ANOVA; Ratio (Test/Reference) of Adjusted Means = 110.17, 90% CI 2-sided [96.05 to 126.37]
Statistical Analysis 3: Comparison: T2DM Normal Renal Function vs T2DM Moderate Renal Impairment; "T2DM Moderate Renal Impairment" was test, "T2DM Normal Renal Function" was reference; Test type: Other — ANOVA; Ratio (Test/Reference) of Adjusted Means = 120.63, 90% CI 2-sided [105.63 to 137.77]
Statistical Analysis 4: Comparison: T2DM Normal Renal Function vs T2DM Severe Renal Impairment; "T2DM Severe Renal Impairment" was test, "T2DM Normal Renal Function" was reference; Test type: Other — ANOVA; Ratio (Test/Reference) of Adjusted Means = 127.06, 90% CI 2-sided [111.26 to 145.12]

5. Secondary Outcome: Maximum Observed Concentration of Unbound Drug (Cmax,u) of Plasma PF-06882961
Description: Cmax,u was defined as maximum observed concentration of unbound drug.
Time Frame: 0 (pre dose), 4 hours (post dose) on Day 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Healthy and Normal Renal Function | T2DM Normal Renal Function | T2DM Mild Renal Impairment | T2DM Moderate Renal Impairment | T2DM Severe Renal Impairment
Number analyzed (Participants) | 8 | 7 | 7 | 8 | 8
ng/mL | 0.5896 (34) | 0.5963 (60) | 0.6662 (32) | 1.055 (25) | 0.7680 (57)

6. Secondary Outcome: Unbound Area Under the Plasma Concentration-Time Profile From Time Zero Extrapolated to Infinite Time (AUCinf,u) of Plasma PF-06882961
Description: AUCinf,u was defined as unbound area under the plasma concentration-time profile from time zero extrapolated to infinite time.
Time Frame: 0 (pre dose), 4 hours (post dose) on Day 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | Healthy and Normal Renal Function | T2DM Normal Renal Function | T2DM Mild Renal Impairment | T2DM Moderate Renal Impairment | T2DM Severe Renal Impairment
Number analyzed (Participants) | 8 | 7 | 6 | 7 | 8
ng*hr/mL | 5.505 (37) | 6.246 (45) | 7.931 (16) | 10.01 (31) | 8.019 (50)

7. Secondary Outcome: Unbound Area Under the Plasma Concentration-Time Profile From Time Zero to the Time of the Last Quantifiable Concentration (AUClast,u) of Plasma PF-06882961
Description: AUClast,u was defined as unbound area under the plasma concentration-time profile from time zero to the time of the last quantifiable concentration.
Time Frame: 0 (pre dose), 4 hours (post dose) on Day 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | Healthy and Normal Renal Function | T2DM Normal Renal Function | T2DM Mild Renal Impairment | T2DM Moderate Renal Impairment | T2DM Severe Renal Impairment
Number analyzed (Participants) | 8 | 7 | 7 | 8 | 8
ng*hr/mL | 5.470 (38) | 6.162 (46) | 7.922 (14) | 10.01 (30) | 7.927 (50)

8. Secondary Outcome: Apparent Clearance (CL/F) of Plasma PF-06882961
Description: Apparent Clearance After Oral Dose (CL/F) was defined as apparent clearance after oral dose on the last day of treatment period.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: liter per hour (L/hr)
Arm/Group | Healthy and Normal Renal Function | T2DM Normal Renal Function | T2DM Mild Renal Impairment | T2DM Moderate Renal Impairment | T2DM Severe Renal Impairment
Number analyzed (Participants) | 8 | 7 | 6 | 7 | 8
liter per hour (L/hr) | 55.17 (30) | 49.32 (49) | 41.08 (19) | 36.83 (48) | 48.93 (46)

9. Secondary Outcome: Apparent Clearance of Unbound Drug After Oral Administration (CLu/F) of Plasma PF-06882961
Description: CLu/F was defined as apparent clearance of unbound drug.
Time Frame: 0 (pre dose), 4 hours (post dose) on Day 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/hr
Arm/Group | Healthy and Normal Renal Function | T2DM Normal Renal Function | T2DM Mild Renal Impairment | T2DM Moderate Renal Impairment | T2DM Severe Renal Impairment
Number analyzed (Participants) | 8 | 7 | 6 | 7 | 8
L/hr | 3631 (37) | 3200 (45) | 2525 (16) | 2000 (31) | 2494 (50)

10. Secondary Outcome: Apparent Volume of Distribution (Vz/F) of Plasma PF-06882961
Description: Vz/F was defined as apparent volume of distribution.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: liter (L)
Arm/Group | Healthy and Normal Renal Function | T2DM Normal Renal Function | T2DM Mild Renal Impairment | T2DM Moderate Renal Impairment | T2DM Severe Renal Impairment
Number analyzed (Participants) | 8 | 7 | 6 | 7 | 8
liter (L) | 600.8 (59) | 552.3 (89) | 372.5 (38) | 438.4 (85) | 565.9 (48)

11. Secondary Outcome: Unbound Vz/F (Vz,u/F) of Plasma PF-06882961
Description: Vz,u/F was defined as apparent volume of distribution of unbound drug.
Time Frame: 0 (pre dose), 4 hours (post dose) on Day 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liter
Arm/Group | Healthy and Normal Renal Function | T2DM Normal Renal Function | T2DM Mild Renal Impairment | T2DM Moderate Renal Impairment | T2DM Severe Renal Impairment
Number analyzed (Participants) | 8 | 7 | 6 | 7 | 8
Liter | 39530 (68) | 35810 (84) | 22890 (30) | 23800 (63) | 28900 (51)

12. Secondary Outcome: Time of Observed Maximum Plasma Concentration (Tmax) of Plasma PF-06882961
Description: Tmax was defined as time to maximum observed concentration. Observed directly from data as time of first occurrence.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Median (Full Range); unit: hour (hr)
Arm/Group | Healthy and Normal Renal Function | T2DM Normal Renal Function | T2DM Mild Renal Impairment | T2DM Moderate Renal Impairment | T2DM Severe Renal Impairment
Number analyzed (Participants) | 8 | 7 | 7 | 8 | 8
hour (hr) | 5.00 [3.00 to 8.00] | 5.00 [5.00 to 8.13] | 6.00 [3.00 to 12.0] | 5.50 [4.00 to 6.00] | 5.00 [4.00 to 6.00]

13. Secondary Outcome: Terminal Elimination Half-Life (T1/2) of Plasma PF-06882961
Description: Plasma terminal elimination half-life (T1/2) is the time measured for the plasma concentration to decrease by one half at the terminal phase.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: hr
Arm/Group | Healthy and Normal Renal Function | T2DM Normal Renal Function | T2DM Mild Renal Impairment | T2DM Moderate Renal Impairment | T2DM Severe Renal Impairment
Number analyzed (Participants) | 8 | 7 | 6 | 7 | 8
hr | 8.111 (3.4828) | 8.139 (2.5640) | 6.640 (2.6551) | 8.907 (4.0497) | 8.058 (0.84962)

14. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs) (All Causalities)
Description: An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. Treatment-emergent adverse event (TEAE) means event between first dose of study treatment and up to 35 days after last dose that were absent before treatment or that worsened relative to pretreatment state. An SAE was an AE resulting in any of death; inpatient hospitalization; life-threatening experience; disability; congenital anomaly or deemed significant for any other reason.
Time Frame: From the first dose of study intervention to the last dose of study treatment date +35 days (up to 13 months)
Population: All participants assigned to study intervention and who took at least 1 dose of study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Healthy and Normal Renal Function | T2DM Normal Renal Function | T2DM Mild Renal Impairment | T2DM Moderate Renal Impairment | T2DM Severe Renal Impairment
Number analyzed (Participants) | 8 | 7 | 8 | 8 | 8
Participants
  Participants with adverse events | 1 | 6 | 1 | 2 | 2
  Participants with serious adverse events | 0 | 0 | 0 | 0 | 0
  Participants with severe adverse events | 0 | 0 | 0 | 0 | 0
  Participants discontinued from study due to adverse events | 0 | 0 | 0 | 0 | 0
  Participants discontinued study drug due to AE and continue Study | 0 | 0 | 0 | 0 | 0
  Participants with dose reduced or temporary discontinuation due to adverse events | 0 | 0 | 0 | 0 | 0

15. Secondary Outcome: Number of Participants With Laboratory Test Abnormalities (Without Regard to Baseline Abnormality)
Description: Laboratory test abnormalities included hematology, chemistry and urinalysis.
Time Frame: From the first dose of study intervention to the last dose of study treatment date +35 days (up to 13 months)
Population: All participants assigned to study intervention and who took at least 1 dose of study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Healthy and Normal Renal Function | T2DM Normal Renal Function | T2DM Mild Renal Impairment | T2DM Moderate Renal Impairment | T2DM Severe Renal Impairment
Number analyzed (Participants) | 8 | 7 | 8 | 8 | 8
Participants
  Hematology: Erythrocytes (10^6/mm^3) < 0.8x LLN: number analyzed (Participants) | 6 | 7 | 8 | 8 | 8
  Hematology: Erythrocytes (10^6/mm^3) < 0.8x LLN | 0 | 0 | 0 | 0 | 1
  Hematology: Ery. Mean Corpuscular HGB Concentration (g/dL) < 0.9x LLN: number analyzed (Participants) | 6 | 7 | 8 | 8 | 8
  Hematology: Ery. Mean Corpuscular HGB Concentration (g/dL) < 0.9x LLN | 0 | 0 | 2 | 0 | 0
  Hematology: Lymphocytes (10^3/mm^3) < 0.8x LLN: number analyzed (Participants) | 5 | 7 | 8 | 8 | 8
  Hematology: Lymphocytes (10^3/mm^3) < 0.8x LLN | 0 | 0 | 0 | 0 | 1
  Hematology: Eosinophils (10^3/mm^3) > 1.2x ULN: number analyzed (Participants) | 5 | 7 | 8 | 8 | 8
  Hematology: Eosinophils (10^3/mm^3) > 1.2x ULN | 0 | 0 | 1 | 1 | 0
  Clinical Chemistry: Bilirubin (mg/dL) > 1.5x ULN | 1 | 0 | 0 | 0 | 0
  Clinical Chemistry: Blood Urea Nitrogen (mg/dL) > 1.3x ULN | 0 | 0 | 4 | 5 | 8
  Clinical Chemistry: Creatinine (mg/dL) > 1.3x ULN | 0 | 0 | 0 | 3 | 8
  Clinical Chemistry: Urate (mg/dL) > 1.2x ULN | 0 | 0 | 1 | 1 | 0
  Clinical Chemistry: Magnesium (mg/dL) < 0.9x LLN: number analyzed (Participants) | 8 | 7 | 7 | 8 | 7
  Clinical Chemistry: Magnesium (mg/dL) < 0.9x LLN | 0 | 0 | 0 | 1 | 0
  Clinical Chemistry: Phosphate (mg/dL) > 1.2x ULN: number analyzed (Participants) | 8 | 7 | 8 | 8 | 7
  Clinical Chemistry: Phosphate (mg/dL) > 1.2x ULN | 0 | 0 | 0 | 0 | 2
  Clinical Chemistry: Bicarbonate (mEq/L) < 0.9x LLN | 0 | 0 | 0 | 0 | 1
  Clinical Chemistry: Glucose (mg/dL) > 1.5x ULN: number analyzed (Participants) | 8 | 7 | 8 | 8 | 7
  Clinical Chemistry: Glucose (mg/dL) > 1.5x ULN | 0 | 4 | 3 | 5 | 3
  Clinical Chemistry: Triacylglycerol Lipase (U/L) > 1.5x ULN | 0 | 2 | 0 | 1 | 2
  Urinalysis: URINE Glucose (Scalar) ≥ 1: number analyzed (Participants) | 8 | 7 | 8 | 8 | 5
  Urinalysis: URINE Glucose (Scalar) ≥ 1 | 0 | 1 | 2 | 2 | 2
  Urinalysis: URINE Protein (Scalar) ≥ 1: number analyzed (Participants) | 8 | 7 | 8 | 8 | 5
  Urinalysis: URINE Protein (Scalar) ≥ 1 | 0 | 0 | 0 | 4 | 4
  Urinalysis: Leukocyte Esterase ≥ 1: number analyzed (Participants) | 8 | 7 | 8 | 8 | 5
  Urinalysis: Leukocyte Esterase ≥ 1 | 0 | 1 | 0 | 0 | 1
  Urinalysis: Hyaline Casts (/LPF) > 1: number analyzed (Participants) | 1 | 1 | 2 | 4 | 5
  Urinalysis: Hyaline Casts (/LPF) > 1 | 0 | 0 | 0 | 0 | 1
  Urinalysis: Bacteria (/HPF) > 20: number analyzed (Participants) | 1 | 1 | 2 | 4 | 5
  Urinalysis: Bacteria (/HPF) > 20 | 1 | 0 | 0 | 0 | 0

16. Secondary Outcome: Number of Participants With Abnormal Vital Signs
Description: The vital signs were measured included pulse rate (beats/min) and blood pressure (mmHg).
Time Frame: From the first dose of study intervention to the last dose of study treatment date +35 days (up to 13 months)
Population: All participants assigned to study intervention and who took at least 1 dose of study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Healthy and Normal Renal Function | T2DM Normal Renal Function | T2DM Mild Renal Impairment | T2DM Moderate Renal Impairment | T2DM Severe Renal Impairment
Number analyzed (Participants) | 8 | 7 | 8 | 8 | 8
Participants
  SITTING SYSTOLIC BLOOD PRESSURE (MMHG): Value < 90mmHg | 0 | 0 | 0 | 0 | 0
  SITTING SYSTOLIC BLOOD PRESSURE (MMHG): Chg ≥ 30mmHg increase | 0 | 0 | 0 | 1 | 1
  SITTING SYSTOLIC BLOOD PRESSURE (MMHG): Chg ≥ 30mmHg decrease | 0 | 0 | 0 | 0 | 1
  SITTING DIASTOLIC BLOOD PRESSURE (MMHG): Value < 50 mmHg | 0 | 0 | 0 | 0 | 0
  SITTING DIASTOLIC BLOOD PRESSURE (MMHG): Chg ≥ 20mmHg increase | 0 | 0 | 1 | 1 | 1
  SITTING DIASTOLIC BLOOD PRESSURE (MMHG): Chg ≥ 20mmHg decrease | 0 | 0 | 0 | 0 | 0
  PULSE RATE (BPM): Value < 40 bpm | 0 | 0 | 0 | 0 | 0
  PULSE RATE (BPM): Value > 120 bpm | 0 | 0 | 0 | 0 | 0

17. Secondary Outcome: Number of Participants With Abnormal Electrocardiograms (ECGs)
Description: ECG parameters included QTCF, PR interval, and QRS interval.
Time Frame: From the first dose of study intervention to the last dose of study treatment date +35 days (up to 13 months)
Population: All participants assigned to study intervention and who took at least 1 dose of study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Healthy and Normal Renal Function | T2DM Normal Renal Function | T2DM Mild Renal Impairment | T2DM Moderate Renal Impairment | T2DM Severe Renal Impairment
Number analyzed (Participants) | 8 | 7 | 8 | 8 | 8
Participants
  PR INTERVAL NOT OTHERWISE SPECIFIED (MSEC): Value ≥ 300: number analyzed (Participants) | 8 | 7 | 8 | 8 | 7
  PR INTERVAL NOT OTHERWISE SPECIFIED (MSEC): Value ≥ 300 | 0 | 0 | 0 | 0 | 0
  PR INTERVAL NOT OTHERWISE SPECIFIED (MSEC): %Chg ≥ 25/50%: number analyzed (Participants) | 8 | 7 | 8 | 8 | 7
  PR INTERVAL NOT OTHERWISE SPECIFIED (MSEC): %Chg ≥ 25/50% | 0 | 0 | 0 | 0 | 0
  QRS INTERVAL NOT OTHERWISE SPECIFIED (MSEC): Value ≥ 140 | 0 | 1 | 0 | 0 | 0
  QRS INTERVAL NOT OTHERWISE SPECIFIED (MSEC): %Chg ≥ 50% | 0 | 0 | 0 | 0 | 0
  QTCF NOT OTHERWISE SPECIFIED (MSEC): 450 < Value ≤ 480 | 0 | 0 | 0 | 1 | 2
  QTCF NOT OTHERWISE SPECIFIED (MSEC): 480 < Value ≤ 500 | 0 | 1 | 0 | 0 | 0
  QTCF NOT OTHERWISE SPECIFIED (MSEC): Value > 500 | 0 | 0 | 0 | 0 | 0
  QTCF NOT OTHERWISE SPECIFIED (MSEC): 30 < Chg ≤ 60 | 0 | 0 | 0 | 0 | 0
  QTCF NOT OTHERWISE SPECIFIED (MSEC): Chg > 60 | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: From the first dose of study intervention to the last dose of study treatment date +35 days (up to 13 months)
Description: The same event may appear as both an adverse event (AE) and an serious adverse event (SAE). An event may be categorized as serious in one participant and as non-serious in another participant, or one participant may have experienced both a serious and non-serious event during the study. Total number at risk below refers to the number of participants evaluable for SAEs or AEs.
Groups:
- Total: Treatment Group Description TBD
Arm/Group | Healthy and Normal Renal Function | T2DM Normal Renal Function | T2DM Mild Renal Impairment | T2DM Moderate Renal Impairment | T2DM Severe Renal Impairment | Total
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/7 | 0/8 | 0/8 | 0/8 | 0/39
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/7 | 0/8 | 0/8 | 0/8 | 0/39
Other Adverse Events (participants affected / at risk) | 1/8 | 6/7 | 1/8 | 2/8 | 2/8 | 12/39
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Healthy and Normal Renal Function (N=8) | T2DM Normal Renal Function (N=7) | T2DM Mild Renal Impairment (N=8) | T2DM Moderate Renal Impairment (N=8) | T2DM Severe Renal Impairment (N=8) | Total (N=39)
Vision blurred (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 1
Constipation (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 0 | 2
Nausea (Gastrointestinal disorders) | 1 | 1 | 0 | 1 | 1 | 4
Fatigue (General disorders) | 0 | 1 | 0 | 0 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 1
Lipase increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 1
SARS-CoV-2 test positive (Investigations) | 0 | 1 | 0 | 0 | 0 | 1
Increased appetite (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 1
Polydipsia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 1
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 1
Polyuria (Renal and urinary disorders) | 0 | 2 | 0 | 0 | 0 | 2
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2020-10-13): https://cdn.clinicaltrials.gov/large-docs/27/NCT04616027/Prot_000.pdf
  • Statistical Analysis Plan (2020-12-10): https://cdn.clinicaltrials.gov/large-docs/27/NCT04616027/SAP_001.pdf